CLINICAL TRIAL: NCT02181088
Title: A Phase Ia Clinical Trial to Assess the Safety and Immunogenicity of New Plasmodium Falciparum Malaria Vaccine Candidates ChAd63 RH5 Alone and With MVA RH5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC057; 2013-005458-31 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: Malaria; Plasmodium falciparum; RH5
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (ChAd63 RH5 low dose) (Experimental): 1 dose of ChAd63 RH5 5 x 10^9 vp intramuscularly
  Interventions: Biological: ChAd63 RH5 low dose
- Group 2A (ChAd63 RH5 full dose) (Experimental): 1 dose of ChAd63 RH5 at 5 x 10^10 vp intramuscularly
  Interventions: Biological: ChAd63 RH5 full dose
- Group 2B (ChAd63 RH5 full dose and MVA RH5 low dose) (Experimental): 1 dose of ChAd63 RH5 at 5 x 10^10 vp intramuscularly and 1 dose MVA RH5 at 1 x 10^8 pfu 8 weeks later intramuscularly
  Interventions: Biological: ChAd63 RH5 full dose; Biological: MVA RH5 low dose
- Group 2C (ChAd63 RH5 full dose and MVA RH5 full dose) (Experimental): 1 dose of ChAd63 RH5 at 5 x 10^10 vp intramuscularly and 1 dose MVA RH5 at 2 x 10^8 pfu 8 weeks later intramuscularly
  Interventions: Biological: ChAd63 RH5 full dose; Biological: MVA RH5 full dose

INTERVENTIONS:
Biological: ChAd63 RH5 low dose — ChAd63 RH5 at 5 x 10^9 vp
  Other Names: ChAd63 RH5
  Arms: Group 1 (ChAd63 RH5 low dose)
Biological: ChAd63 RH5 full dose — ChAd63 RH5 at 5 x 10^10 vp
  Other Names: ChAd63 RH5
  Arms: Group 2A (ChAd63 RH5 full dose); Group 2B (ChAd63 RH5 full dose and MVA RH5 low dose); Group 2C (ChAd63 RH5 full dose and MVA RH5 full dose)
Biological: MVA RH5 low dose — MVA RH5 at 1 x 10^8 pfu
  Other Names: MVA RH5
  Arms: Group 2B (ChAd63 RH5 full dose and MVA RH5 low dose)
Biological: MVA RH5 full dose — MVA RH5 at 2 x 10^8 pfu
  Other Names: MVA RH5
  Arms: Group 2C (ChAd63 RH5 full dose and MVA RH5 full dose)

SUMMARY:
The purpose of this study is to assess two new malaria vaccines, ChAd63 RH5 and MVA RH5, at different doses and alone or in combination. The study will enable us to assess the safety of the vaccines and the extent of the immune response in healthy volunteers. We will do this by giving volunteers one or two vaccinations, doing blood tests and collecting information about any symptoms that occur after vaccination. This is the first trial to use these vaccines in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including human immunodeficiency virus (HIV) infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* History of clinical malaria (any species)
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's general practitioner (GP) to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety of ChAd63 RH5 when administered alone and in heterologous prime-boost with MVA RH5 | 240 days
  Occurrence of solicited and unsolicited adverse events will be monitored at each clinic visit from diary cards, clinical review, clinical examination (including observations) and laboratory results.

SECONDARY OUTCOMES:
To assess the cellular and humoral immunogenicity of ChAd63 RH5 when administered alone, and in heterologous prime-boost with MVA RH5 in healthy volunteers. | 240 days
  P. falciparum RH5-specific immunogenicity will be assessed by a variety of immunological assays. These may include ex vivo ELISpot assays for interferon gamma and flow cytometry assays, as well as antibody ELISAs, functional antibody assays and B cell analyses. Other exploratory immunological assays including cytokine analysis, other antibody assays, anti-adenovirus antibodies, DNA analysis of genetic polymorphisms potentially relevant to vaccine immunogenicity and gene expression studies amongst others may be performed at the discretion of the Investigators.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford
  - Wellcome Trust CRF, Southampton General Hospital, University of Southampton, Southampton